CLINICAL TRIAL: NCT00680576
Title: Adolescent Substance Abuse: Progressive Treatment
Acronym: ADAPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DA023568; R01DA023568 (NIH)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Substance Abuse
Keywords: adolescent substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Eight weeks of individual CBT for adolescents who have completed six weeks of group therapy and continue to use drugs.
  Interventions: Behavioral: CBT, Cognitive Behavioral Therapy
- 2 (Active Comparator): Eight weeks of FFT for adolescents who have received six weeks of group therapy and continue to use drugs.
  Interventions: Behavioral: FFT, Family Functional Therapy

INTERVENTIONS:
Behavioral: CBT, Cognitive Behavioral Therapy — Eight weekly sessions of individual Cognitive Behavioral Therapy, to develop skills enabling adolescents stop or reduce their drug use.
  Arms: 1
Behavioral: FFT, Family Functional Therapy — Eight weekly sessions of Functional Family Therapy designed to strengthen family relationships and build skills to help the adolescent stop or reduce his/her drug use.
  Arms: 2

SUMMARY:
The purpose of this study is to find out more about how to provide effective further treatment for adolescents who have received six weeks of group therapy for substance-use problems and continue to use drugs. Treatments used in the study include a group therapy (MET/CBT), an individual therapy (CBT), and a family therapy (FFT). The study will look at whether abstinence or a very low level of use is a better guide for deciding whether further treatment is needed, how well different combinations of treatment work to reduce substance use, and whether it is possible to predict in advance which adolescents will respond best to which types of treatment. Study investigators expect that a treatment strategy using what is learned about these issues in the first half of the project to develop an "adaptive" treatment model will work better than a "fixed" treatment to reduce adolescent substance use.

ELIGIBILITY:
Inclusion Criteria:

1. 13 to 18 years if age
2. Meet DSM-IV (APA, 1994) diagnostic criteria for substance abuse or dependence
3. Live in the Albuquerque metropolitan area or surrounding communities
4. Sufficient residential stability to permit probable contact at follow-up (e.g., not homeless at time of intake).

Exclusion Criteria:

1. There is evidence of psychotic or organic state of sufficient severity to interfere with the understanding of study instruments and procedures
2. The adolescent is deemed dangerous to self or others during evaluation
3. Services other than outpatient treatment are required for the adolescent (e.g., inpatient, detoxification)
4. Marijuana use is reported as being less than 13% of days in the previous 90 days.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2008-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Urine drug screens | Pretx, 6, 14 and 22 weeks, 3 and 6 months after initial treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Holly B Waldron, Ph.D., Principal Investigator — Oregon Research Institute Center for Family and Adolescent Research (ORI/CFAR)
Locations (1):
- Oregon Res. Inst. Center for Family & Adolescent Research (CFAR), Albuquerque, New Mexico, United States